CLINICAL TRIAL: NCT05495750
Title: The Impact of Adding Ultrasound Guided Bilateral Suprazygomatic Maxillary Nerve Block to General Anesthesia on Systemic Inflammatory Response in Cleft Palate Surgeries ; A Randomized Control Trial
Brief Title: Suprazygomatic Maxillary Nerve Block Effect on Systemic Inflammatory Response in Cleft Palate Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alaa Mohamed Abdel Salam Ibrahim Soliman (Other)
Responsible Party: Sponsor-Investigator, Alaa Mohamed Abdel Salam Ibrahim Soliman, Assistant Lecturer, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MD 141/2022
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Perioperative Inflammatory Response; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxillary block group (Active Comparator): The ultrasound probe will be placed in the infra zygomatic area, with an inclination of 45 degrees in the transverse plane. A 27-gauge 38-mm needle will be used for the injection. The needle will be inserted perpendicular to the skin at the frontozygomatic angle and advanced to the greater wing of the sphenoid. The needle will be then redirected and advanced to the pterygopalatine fossa.
  Loss of resistance after passing through the temporalis muscle will assist in determining the puncture depth, and real-time ultrasound guidance will allow seeing the spread of local anesthetic in the pterygopalatine fossa.
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- Control group (No Intervention): Patients will receive only general anesthesia with regulated doses of IV opioids.

INTERVENTIONS:
Drug: Bupivacaine 0.25% Injectable Solution — ultrasound-guided bilateral suprazygomatic maxillary nerve block using 0.15 ml/kg.
  Other Names: supra zygomatic maxillary nerve block
  Arms: Maxillary block group

SUMMARY:
the aim is to determine the value of adding bilateral supra zygomatic maxillary nerve block to general anesthesia in attenuating the systemic inflammatory response in paediatrics.

DETAILED DESCRIPTION:
Cleft lip and palate are some of the most common craniofacial malformations, with an incidence ranging between 0.1 and 1.1 per 1000 births. Early surgical intervention for cleft palate (CP) repair is essential for proper feeding and phonation as well as reduction of complications such as frequent sinusitis and other respiratory tract infections.

Surgical injury stimulates the systemic inflammatory response. The neuroendocrine response leads to stimulation of the sympathetic nervous system resulting in tachycardia, hypertension and activation of the hypothalamic-pituitary adrenal axis. This induces the release of hormones such as adrenocorticotropic hormone (ACTH), catechol-amines (norepinephrine and epinephrine) and cortisol and increase in white cell count which is proposed to have a detrimental effect on the postoperative immunity. Furthermore, the production of pro-inflammatory cytokines including interleukins (IL) e.g.IL-1, IL-6, IL-8 and tumour necrosis factor alpha (TNF-α) by innate immune cells such as neutrophils and macrophages, interacting with damaged cells and platelets, leads to the production of acute phase proteins from the liver such as C-reactive protein (CRP), fibrinogen and complement proteins.

Regional blocks provide good pre-emptive analgesia when given in combination with general anaesthesia (GA). It is associated with hemodynamic stability, rapid recovery, reduction of supplemental analgesia consumption in addition to favourable effect on systematic inflammatory response. Using bilateral suprazygomatic approach of maxillary nerve block during CP repair is hypothesized to provide such mentioned settlement of a regional block.

ELIGIBILITY:
Inclusion Criteria:

* Primary and secondary cleft palate Surgeries.
* American Society of Anesthesiologists physical status (ASA) I to II patients.
* Age group: 1-5 years old.

Exclusion Criteria:

* Presence of coagulation disorders.
* Peripheral neuropathy.
* Local infection or lesion in puncture site.
* Allergy to local Anesthetics.
* Physical status: ASA III or above.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Interleukin 6 serum level. | 3-5 hours
  Two blood samples will be withdrawn in both groups, the first sample immediately after induction of general anaesthesia, endotracheal tube insertion and the other sample will be withdrawn after completion of surgery and before recovery of the patient

SECONDARY OUTCOMES:
Serum Cortisol level | 3-5 hours
  Two blood samples will be withdrawn in the both groups, the first sample immediately after induction of general anaesthesia, endotracheal tube insertion and the other sample will be withdrawn after completion of surgery and before recovery of the patient
Plasma glucose level | 3-5 hours
  Two blood samples will be withdrawn in the both groups, the first sample immediately after induction of general anaesthesia, endotracheal tube insertion and the other sample will be withdrawn after completion of surgery and before recovery of the patient
C-Reactive protein (CRP) | 3-5 hours
  Two blood samples will be withdrawn in the both groups, the first sample immediately after induction of general anaesthesia, endotracheal tube insertion and the other sample will be withdrawn after completion of surgery and before recovery of the patient
Total leucocytic count | 3-5 hours
  Two blood samples will be withdrawn in the both groups, the first sample immediately after induction of general anaesthesia, endotracheal tube insertion and the other sample will be withdrawn after completion of surgery and before recovery of the patient
CHIPPS score | 1 hour (h), 2 h, 4 h, 6 h, 8 h, 12 h postoperatively.
  Score 0 , Score 1 , Score 2
The number of rescue analgesia doses postoperatively | 12 hours postoperative
  IM Diclofenac(0.5 mg/kg) will be given as rescue analgesia for patients if CHIPPS was > 3/10
time needed till the need of first dose recorded of rescue analgesia | 12 hours post operative
  IM Diclofenac(0.5 mg/kg) will be given as rescue analgesia for patients if CHIPPS was > 3/10
Time needed to start oral feeding will be recorded | 12 hours postoperative
  time of starting oral feeding

CONTACTS AND LOCATIONS:
Overall Officials: Sherif S Sultan, MD, Study Director — Ainshams University; Tamer N Ibrahim AbdelRahman, MD, Study Chair — Ainshams Univeristy; Sohib M Galal, MD, Study Chair — Ainshams Univeristy; Sarah A Salem, MD, Study Chair — Ainshams Univeristy
Locations (1):
- Faculty of dentisry Ainshams univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Summary results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: Internet search by keywords